CLINICAL TRIAL: NCT04393389
Title: All Comers Post Market Clinical Follow-up to Continue the Surveillance of the Acotec Drug Coated PTA Catheter Orchid, Tulip and Litos in Lower Limb Treatment
Brief Title: Acotec DCB Post Market Clinical Follow-up
Acronym: FLOWER
Status: Recruiting | Type: Observational
Sponsor: Acotec Scientific Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Acotec-07
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-CLI group: Rutherford Clinical Category (RCC) 2-3
  Interventions: Device: AcoArt Orchid (0.035"), AcoArt Tulip (0.018") and AcoArt Litos (0.014") percutaneous transluminal angioplasty (PTA) paclitaxel drug coated balloon catheter manufactured by Acotec Scientific Co., Ltd.
- CLI group: critical limb ischemia，Rutherford Clinical Category (RCC) 4-6
  Interventions: Device: AcoArt Orchid (0.035"), AcoArt Tulip (0.018") and AcoArt Litos (0.014") percutaneous transluminal angioplasty (PTA) paclitaxel drug coated balloon catheter manufactured by Acotec Scientific Co., Ltd.

INTERVENTIONS:
Device: AcoArt Orchid (0.035"), AcoArt Tulip (0.018") and AcoArt Litos (0.014") percutaneous transluminal angioplasty (PTA) paclitaxel drug coated balloon catheter manufactured by Acotec Scientific Co., Ltd. — All comers Post Market Clinical Follow-up to continue the surveillance of the Acotec Drug Coated PTA Catheter AcoArt Orchid, AcoArt Tulip and AcoArt Litos in lower limb treatment

SUMMARY:
All-comers, prospective, multi-center, single-arm, non-interventional post market clinical follow-up (PMCF) Cohort 1 - Claudicants: Rutherford Clinical Category (RCC) 2-3 Cohort 2 - Critical Limb Ischemia: Rutherford Clinical Category (RCC) 4-6

DETAILED DESCRIPTION:
To prospectively collect and assess safety and efficacy data on the AcoArt drug-coated PTA balloon catheters carrying the CE Mark per current Instructions for Use in a real-world cohort of patients with symptomatic arterial disease undergoing endovascular lower limb revascularization per the institution's standard practice.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient is ≥ 18 years old at the time of consent.
* 2. Significant stenosis (≥70%) or occlusions of de-novo or restenotic lesion(s) located in iliac, superficial femoral, popliteal and/or infra-popliteal arteries suitable for angioplasty per operator visual assessment.
* 3. Lesion(s) can be treated with available AcoArt Orchid (0.035"), AcoArt Tulip (0.018") and AcoArt Litos (0.014") DCB device per current IFU.
* 4. Subject has provided written informed consent prior to participation in the PMCF, understands the purpose of this PMCF and agrees to comply with all protocol-specified examinations and follow-up appointments.
* 5. Rutherford Classification Category 2-6 Subjects with Rutherford Category 2 have gone through a conservative therapy without success.
* 6. Inflow lesion treated prior to target lesion treatment

Exclusion Criteria:

* 1. Rutherford Classification Category 0, 1
* 2. Patient already enrolled in other investigational (interventional) studies that would interfere with study endpoints
* 3. Inability to tolerate required antithrombotic or antiplatelet therapies.
* 4. Non-dilatable severely calcified lesion.
* 5. Known hypersensitivity/allergy to components of the investigational device
* 6. Un-treated acute or subacute thrombus in the target lesion.
* 7. Life expectancy < 1 year.
* 8. Pregnancy or female patient with child bearing potential not taking adequate contraceptives or currently lactating.
* 9. Other comorbidities, which in the opinion of the investigator limit longevity or likelihood of compliance with protocol follow up.
* 10. Myocardial infarction or stroke within 30 days prior to index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with symptomatic arterial disease undergoing endovascular lower limb revascularization per the institution's standard practice.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint - non-CLI group | 12 Months
  Freedom from clinically-driven target lesion revascularization (CD-TLR) within 12 months after index procedure, which is defined as any re-intervention within the target lesion(s) due to recurrent clinical symptoms of PAD (increase of one Rutherford class or more) and/or drop of ankle-brachial index (≥20% or >0.15 when compared with maximum early post-procedural level).
Primary efficacy endpoint -CLI group | 6 Months
  Freedom from clinically-driven TLR within 6 months after index procedure, which is defined as any re-intervention within the target lesion(s) due to delayed or worsening wound healing, new or recurrent wound, or worsening Rutherford class.
Primary safety endpoint- non-CLI group | 30 days
  A composite of freedom from major adverse limb events and perioperative death (MALE-POD) through 30 days after index procedure. A major adverse limb event is defined as above-ankle amputation or major reintervention (ie, new bypass graft, major surgical graft revision such as a jump graft or an interposition graft, or thrombectomy/thrombolysis) of the treated limb.
Primary safety endpoint- CLI group | 12 Months
  A composite of freedom from device- and procedure-related mortality, freedom from major target limb amputation and TLR within 12 months post-index procedure

SECONDARY OUTCOMES:
Rate of Any TLR (including clinically-driven and incidental TLR) | 6 months,12 months,24 months, 36months,48 months,60 months
  Any TLR (including clinically-driven and incidental TLR) at 6,12, 24, 36, 48, 60 months post-procedure
Rate of Target vessel revascularization (TVR) | 6 months,12 months,24 months, 36months,48 months,60 months
  Target vessel revascularization (TVR) at 6, 12, 24, 36, 48, 60 months post-procedure
Rate of Target limb revascularization | 6 months,12 months,24 months, 36months,48 months,60 months
  Target limb revascularization at 6, 12, 24, 36, 48, 60 months post-procedure
Rate of CD-TLR | 6 months,12 months,24 months, 36months,48 months,60 months
  CD-TLR at 6, 24, 36, 48, 60 months post-procedure
Rate of All-cause mortality | 6 months,12 months,24 months, 36months,48 months,60months
  All-cause mortality at 6, 12, 24, 36, 48, 60 months post procedure
Rate of Device- or procedure-related death | 30 days, 6 months
  Device- or procedure-related death at 30 days and 6 months
Rate of Major amputation | 6 months,12 months,24 months, 36months,48 months,60 months
  Major amputation at 6, 12, 24, 36, 48, 60 months post procedure
Rate of Technical success | Post procedure
  Technical success defined as final in-lesion residual diameter stenosis ≤50% by angiographic visual estimate at the end of the index procedure without device malfunction.
Rate of Procedural success | Post procedure
  Procedural success defined as technical success without procedural complications (death, major target limb amputation, thrombosis of the target lesion, or CD-TLR) prior to discharge
Change in Rutherford clinical category (target limb) | 6 months,12 months,24 months, 36months,48 months,60 months
  Changes in Rutherford clinical category (target limb) at 6, 12, 24, 36, 48, 60 months post-procedure compared to baseline
Rate of primary sustained clinical improvement | 6 months,12 months,24 months, 36months,48 months,60 months
  Primary sustained clinical improvement, defined as improvement in Rutherford classification by one or more categories compared with baseline, without TLR.
Rate of secondary sustained clinical improvement | 6 months,12 months,24 months, 36months,48 months,60 months
  Secondary sustained clinical improvement, defined as improvement in Rutherford classification by one or more categories compared with baseline, including patients with TLR
Rate of (Major) Amputation-free survival - CLI group | 6 months,12 months,24 months, 36months,48 months,60 months
  (Major) Amputation-free survival at 6, 12, 24, 36, 48, 60 months post-procedure
Rate of Minor amputation - CLI group | 6 months,12 months,24 months, 36months,48 months,60 months
  Minor amputation at 6, 12, 24, 36, 48, 60 months post-procedure
Rate of Wound healing - CLI group | 60 months
  healed or not; if not, improving, stagnant,worsening
New or recurrent wound of the target limb - CLI group | 60 months
  New or recurrent wound of the target limb

CONTACTS AND LOCATIONS:
Overall Officials: Schmidt Andrej, Principal Investigator — Department of Angiology, University Hospital Leipzig
Locations (7):
- Germany (7):
  - Halle, Halle, Saxony-Anhalt
  - Eilenburg, Eilenburg
  - Department of Angiology, University Hospital Leipzig,, Leipzig
  - Elblandklinikum Radebeul, Radebeul
  - Elblandklinikum Radebeul, Riesa
  - REGIOMED Klinikum Sonneberg, Sonneberg
  - KKH Torgau, Torgau